CLINICAL TRIAL: NCT05139901
Title: Usefulness of DORNASE (Pulmozyme®) in Patients With COVID-19 Respiratory Insufficiency on High-Flow Oxygen Therapy
Brief Title: Usefulness of DORNASE in COVID-19 on HFNO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the Omicron version of SARS-CoV-2 the COVID-pneumonia patients ran out
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Marko Zlicar, Head of department, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DTS_pulmosyme
Record Dates: First submitted 2021-11-30; First posted 2021-12-01 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — dornase alfa; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blind randomised
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4% saline (Active Comparator): 4% Saline inhalations twice daily
  Interventions: Drug: Saline
- Pulmosyme (Experimental): DNAse alpha inhalations twice daily
  Interventions: Drug: Dornase Alfa

INTERVENTIONS:
Drug: Dornase Alfa — inhalations twice daily
  Arms: Pulmosyme
Drug: Saline — inhalations twice daily
  Other Names: 4% Saline
  Arms: 4% saline

SUMMARY:
COVID-19 pneumonia manifests among others with a thick bronhial secretion. It contains an increased number of neutrophil extracellular traps (NETs), formed during netosis. DNA is a major component in NETs. DNAse alfa (Pulmozyme®, Roche) is a recombinant human enzyme, registered for inhalations in patients with Cystic fibrosis, in which NETs are also a typical characteristic. DNAse alfa inhalations are typically well tolerated and with no major side effects. Some initial reports exist of using DNAse alfa inhalations in COVID-19 patients, that had benefitial effects. There are some trials registered with ClinicalTrials, investigating the usufulness of DNAse alfa in intubated patients, but the investigators have no knowledge of a trial, investigating the usufulness of this drug in patients receiving High Flow Nasal Oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 RNA PCR swab
* inflamatory phase of infection
* HFNO

Exclusion Criteria:

* pregnancy
* previous treatment with DNAse alfa

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Intubations | 7 days
  Number of intubations necessary

SECONDARY OUTCOMES:
PaO2/FiO2 | 7 days
  Increase in PaO2/FiO2 ratio
inflamation | 7 days
  Reduction of inflamation

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided